CLINICAL TRIAL: NCT01672216
Title: Triple Target Treatment (3T) Combining Amplitude Modulated Middle Frequency (AM-MF) Stimulation With Electromyography (EMG)EMG-Biofeedback Versus EMG-Biofeedback in Chronic Obstipation
Brief Title: Multicenter Randomized Controlled Trial to Compare the Outcome of Conservative Triple Target Treatment With EMG-Biofeedback in Chronic Obstipation
Acronym: 3T-CO
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: dr. schwandner (Other)
Responsible Party: Sponsor-Investigator, dr. schwandner, Head of Coloproctology, University of Giessen
Organization: University of Giessen (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 101/12 ethics comm. Giessen
Record Dates: First submitted 2012-08-07; First posted 2012-08-24 (Estimated); Last update posted 2013-09-23 (Estimated); Status verified 2013-09

CONDITIONS: Chronic Obstipation
Keywords: Exercise Therapy; Biofeedback (Psychology); Adult; Chronic Obstipation/*therapy; EMG - Biofeedback; EMG - Triggered Stimulation; Augmented biofeedback

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Triple Target Treatment (Experimental): In the 3T arm, patients were stimulated with a carrier wave of 25 KHz and biphasic modulations of the pulse train of 40 Hz. Anxious patients trained at first only in the biofeedback mode. The stimulation was introduced after four weeks for these patients. Patients were instructed to carry out the training at home, with an alternating combination in the morning and with EMG-triggered stimulation in the evening, each for 20-minute periods. Apart from this, the protocol of the active treatment group was identical to that of the control group.
  Interventions: Device: Combination of EMG-biofeedback plus EMG-triggered AM-MF-stimulation
- EMG-biofeedback alone (Active Comparator): In the biofeedback arm, patients were instructed to carry out EMG-biofeedback training at home, standing, mornings and evenings, for 20-minute periods. The core of the task was to pull the plug-electrode upward inside the anal channel, like a lift, and to hold it there during varying periods of tension. This can only be done successfully if the perineum rises and at the same time the puborectal muscle is activated. Just squeezing the sphincter muscles does not produce this lifting effect.
  Interventions: Device: EMG-biofeedback alone

INTERVENTIONS:
Device: Combination of EMG-biofeedback plus EMG-triggered AM-MF-stimulation
  Arms: Triple Target Treatment
Device: EMG-biofeedback alone
  Arms: EMG-biofeedback alone

SUMMARY:
Previous studies revealed only a low evidence for the various biofeedback methods and pelvic floor exercises for treatment of chronic obstipation. The number of randomized controlled trials is low with in part significant systemic deficiencies. However, the results from the previous study with 3T treatment in patients with obstructed defecation syndrome (ODS) are so promising that a further randomized controlled trial appears useful to demonstrate a higher degree of evidence. The purpose of this study is to determine whether triple target treatment (3T) or EMG-Biofeedback alone are effective in the treatment of chronic obstipation and if the duration of treatment (3, 6 or 9 months) influence the efficacy.

DETAILED DESCRIPTION:
Methods in this parallel-group randomized multicenter study with blinded observer we enroll 140 patients with chronic obstipation. The study is divided into two trials. After three months the first trial is completed and can be extended directly into the second trial (completed after 12 months) after an interim analysis. Primary endpoints are changes from baseline to three and twelve months in the Altomare ODS Score.

ELIGIBILITY:
Inclusion Criteria:

* All Patients with chronic obstipation (Rom criteria II)

Exclusion Criteria:

* Chronic inflammatory bowel disease, systemic peripheral neuropathy (MS, diabetes), disorders of enteric nervous system (Hirschsprung disease, chagas, IND, myopathy desmosis coli), idiopathic megacolon/megarectum, patients with mental or intellectual deficits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2012-08; Primary Completion 2014-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Altomare ODS Score in its validated form after 3 and 12 months, compared to baseline. | 3 months

SECONDARY OUTCOMES:
Constipation severity instrument (CSI) in adapted German form after 3 and 12 months, compared to baseline. | 3 and 12 months
Modified Wexner Incontinence Score after 3 and 12 months, compared to baseline | 3 and 12 Months
Patient Assessment of Constipation Quality of Life Questionnaire (PAC-QoL) after 3 and 12 months compared to baseline, as well as between the two treatment groups over the course of time as compared to baseline. | 3 and 12 months
Hinton Test after 3 and 12 months | 3 and 12 months
Cleveland Clinic Incontinence Score (CCS) in its validated German form after 3 and 12 months, compared to baseline | 3 and 12 months
Adapted Vaizey score after 3 and 12 months compared to baseline | 3 and 12 months
International Consultation on Incontinence Questionnaire Short Form (ICIQ-SF) applied to patients with urine incontinence after 3 and 12 months, compared to baseline. | 3 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Thilo Schwandner, Dr., Principal Investigator — University of Giessen
Locations (1):
- University of Gießen, Dept. of General Surgery, Giessen, Hesse, Germany

REFERENCES:
- [Background] Schwandner T, Hecker A, Hirschburger M, Hecker M, Kierer W, Padberg W. Does the STARR procedure change the pelvic floor: a preoperative and postoperative study with dynamic pelvic floor MRI. Dis Colon Rectum. 2011 Apr;54(4):412-7. doi: 10.1007/DCR.0b013e318205ddda. PMID 21383560